CLINICAL TRIAL: NCT00634634
Title: Phase I/II Trial of Letrozole (Femara) and Sorafenib (Nexavar) in Postmenopausal Women With Hormone-Receptor Positive Locally Advanced or Metastatic Breast Cancer
Brief Title: Phase I/II Trial of Letrozole and Sorafenib in Post-Menopausal Hormone-Receptor + Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH); Bayer (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Deborah Toppmeyer, MD, Professor of Medicine, Chief Medical Officer, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040706; NJ 1107 (Other: CINJOG); 0220070284 (Other: IRB #); NCI-2012-00525 (Other: NCI #); 0220070284 (Other: Rutgers Cancer Institute of New Jersey); Pro2018001861 (Other: Rutgers IRB#)
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer; Postmenopausal Women with Hormone Receptor-Positive Locally Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib and Letrozole (Experimental)
  Interventions: Drug: Sorafenib; Drug: Letrozole

INTERVENTIONS:
Drug: Sorafenib — sorafenib dose will be given at a daily dose to be determined based upon the phase of study that patient is enrolled The phase II dose of sorafenib will be determined from the phase I portion of the study.
  Other Names: Nexavar
Drug: Letrozole — Patients will take letrozole orally at a daily dose of 2.5 mg/day on Days 1 through 28
  Other Names: Femara

SUMMARY:
Letrozole is an aromatase inhibitor that is approved in the first-line treatment of postmenopausal women with hormone receptor-positive or hormone receptor unknown locally advanced or metastatic breast cancer. Sorafenib may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth. This phase I/II trial is studying the side effects and best dose of sorafenib when given in combination with letrozole and to see how well they work in treating postmenopausal women with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed invasive breast cancer
2. Stage IIIB, IIIC with T4 lesion or Stage IV disease
3. Breast cancer must be ER-positive and/or PR-positive
4. Age ³ 18 years of age
5. ECOG performance status 0, 1 or 2
6. Able to swallow and oral medication
7. Adequate end organ function
8. Written informed consent

Exclusion Criteria:

1. Prior hormonal therapy for metastatic disease
2. Prior chemotherapy for metastatic disease
3. Prior treatment with sorafenib
4. Brain metastases or leptomeningeal disease
5. Evidence or history of bleeding
6. Thrombolic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-08-11 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2023-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Tan, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (4):
- United States (4):
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Cooper Hospital/University Medical Center, Voorhees Township, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 13 participants in Phase I + 39 participants enrolled in Phase II = 52 participants that appear to be enrolled in this study.
Groups:
- Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level -1: Sorafenib: sorafenib dose will be given at a daily dose to be determined based upon the phase of study that patient is enrolled The phase II dose of sorafenib will be determined from the phase I portion of the study.
  Dose Level -1: Sorafenib 400mg po every other day. Letrozole: Patients will take letrozole orally at a daily dose of 2.5 mg/day on Days 1 through 28
- Phase l Sorafenib Dose Escalation and Letrozole 2.5mg Daily Dose Level 0:Sorafenib 400mg 1X Daily: Sorafenib: s dose will be given at a daily dose to be determined based upon the phase of study that patient is enrolled The phase II dose of sorafenib will be determined from the phase I portion of the study
  Dose Level 0: Sorafenib 400mg 1X daily Letrozole: Patients will take letrozole orally at a daily dose of 2.5 mg/day on Days 1 through 28
- Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level 1: Sorafenib 400mg 2X Day: Sorafenib: sorafenib dose will be given at a daily dose to be determined based upon the phase of study that patient is enrolled The phase II dose of sorafenib will be determined from the phase I portion of the study.
  Dose Level 1: Sorafenib 400mg 2X day. Letrozole: Patients will take letrozole orally at a daily dose of 2.5 mg/day on Days 1 through 28
- Phase II Arm - Sorafenib at MTD (400mg) 2x a Day + Letrozole 2.5 mg po Daily: Sorafenib 400mg 2X day. Letrozole: Patients will take letrozole orally at a daily dose of 2.5 mg/day
Period: Overall Study
Arm/Group | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level -1 | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg Daily Dose Level 0:Sorafenib 400mg 1X Daily | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level 1: Sorafenib 400mg 2X Day | Phase II Arm - Sorafenib at MTD (400mg) 2x a Day + Letrozole 2.5 mg po Daily
Started | 1 | 3 | 9 | 39
Completed | 1 | 3 | 9 | 39
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level -1 | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg Daily Dose Level 0:Sorafenib 400mg 1X Daily | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level 1: Sorafenib 400mg 2X Day | Phase II Arm - Sorafenib at MTD (400mg) 2x a Day + Letrozole 2.5 mg po Daily | Total
Number analyzed (Participants) | 1 | 3 | 9 | 39 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 4 | 36 | 40
  >=65 years | 1 | 3 | 5 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 9 | 39 | 52
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 10 | 10
  White | 1 | 3 | 9 | 25 | 38
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 9 | 39 | 52

OUTCOME MEASURES:

1. Primary Outcome: Sorafenib in Combination With Fixed Dose of of 2.5mg of Letrozole Maximum Tolerated Dose (MTD)
Description: The highest dose of the drug that does not cause unacceptable side effects. The maximum tolerated dose be testing increasing doses until the highest dose with acceptable side effects is found.
Time Frame: twenty eight days
Population: The primary outcome is the maximum tolerated dose, which is the highest dose of the drug that does not cause unacceptable side effects. The maximum tolerated dose was only analyzed. Then phase 2 added 39 participates.
Measure: Number; unit: milligrams twice daily
Groups:
- Sorafenib in Combination With Fixed Dose of of 2.5mg of Letrozole Maximum Tolerated Dose (MTD): The highest dose of the drug that does not cause unacceptable side effects. The maximum tolerated dose be testing increasing doses until the highest dose with acceptable side effects is found.
Arm/Group | Sorafenib in Combination With Fixed Dose of of 2.5mg of Letrozole Maximum Tolerated Dose (MTD)
Number analyzed (Participants) | 13
milligrams twice daily | 400

2. Secondary Outcome: Clinical Benefit Rate Using the Response Evaluation Criteria in Solid Tumors (RECIST) Guidelines (Version 1.1) to Letrozole and Sorafenib
Description: Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the malignant lymph nodes are used for tumor measurements. Included will be: complete response, partial response or stable disease of letrozole and sorafenib in the treatment of postmenopausal participants with hormone receptor- positive locally advanced or metastatic breast cancer.
  Clinical Benefit Rate (CBR) = Progressive Free (PF) + Stable Disease (SD)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level -1 | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg Daily Dose Level 0:Sorafenib 400mg 1X Daily | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level 1: Sorafenib 400mg 2X Day | Phase II Arm - Sorafenib at MTD (400mg) 2x a Day + Letrozole 2.5 mg po Daily
Number analyzed (Participants) | 1 | 3 | 9 | 39
Participants | 0 | 3 | 4 | 23

3. Secondary Outcome: Median Progressive-Free Survival (PFS)
Description: PFS based on the Kaplan-Meier method is defined as the time between randomization and documented disease progression (PD) per RECIST 1,0 criteria or death, or is censored at time of last disease assessment. Per RECIST 1.0f or target lesions, PD is at least a 20% increase in sum LD of target lesions, taken as reference the smallest sum LD recorded at treatment started. Based on the time between the first day of treatment and and the date of disease progression.
Time Frame: Approximately 4.6 years
Measure: Median (Full Range); unit: months
Arm/Group | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level -1 | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg Daily Dose Level 0:Sorafenib 400mg 1X Daily | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level 1: Sorafenib 400mg 2X Day | Phase II Arm - Sorafenib at MTD (400mg) 2x a Day + Letrozole 2.5 mg po Daily
Number analyzed (Participants) | 1 | 3 | 9 | 39
months | 0 [0 to 0] | 10 [5 to 15] | 34.5 [5 to 66] | 11 [1 to 52]

4. Secondary Outcome: Overall Survival (OS) Assessed as Mean Months
Description: From the start of treatment to the end of the study (three years) that participants are still alive. Measured by the mean number.
Time Frame: Approximately 4.6 years
Measure: Mean (Full Range); unit: months
Arm/Group | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level -1 | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg Daily Dose Level 0:Sorafenib 400mg 1X Daily | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level 1: Sorafenib 400mg 2X Day | Phase II Arm - Sorafenib at MTD (400mg) 2x a Day + Letrozole 2.5 mg po Daily
Number analyzed (Participants) | 1 | 3 | 9 | 39
months | 44 [44 to 44] | 21 [17 to 25] | 49.6 [38 to 56] | 24.8 [1 to 49]

ADVERSE EVENTS:
Time Frame: Approximately 4.6 years
Arm/Group | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level -1 | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg Daily Dose Level 0:Sorafenib 400mg 1X Daily | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level 1: Sorafenib 400mg 2X Day | Phase II Arm - Sorafenib at MTD (400mg) 2x a Day + Letrozole 2.5 mg po Daily
All-Cause Mortality (participants affected / at risk) | 1/1 | 2/3 | 7/9 | 24/39
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/3 | 0/9 | 3/39
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3 | 9/9 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level -1 (N=1) | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg Daily Dose Level 0:Sorafenib 400mg 1X Daily (N=3) | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level 1: Sorafenib 400mg 2X Day (N=9) | Phase II Arm - Sorafenib at MTD (400mg) 2x a Day + Letrozole 2.5 mg po Daily (N=39)
Hypertension (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatobiliary (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Headaches (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level -1 (N=1) | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg Daily Dose Level 0:Sorafenib 400mg 1X Daily (N=3) | Phase l Sorafenib Dose Escalation and Letrozole 2.5mg po Daily Dose Level 1: Sorafenib 400mg 2X Day (N=9) | Phase II Arm - Sorafenib at MTD (400mg) 2x a Day + Letrozole 2.5 mg po Daily (N=39)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 7 (11) | 28 (67)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (8) | 11 (14)
Vascular (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 15 (23)
General (General disorders) | 0 (0) | 0 (0) | 3 (7) | 19 (64)
Blood (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (12)
Reproductive (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (10) | 19 (39)
Pain (General disorders) | 0 (0) | 0 (0) | 4 (8) | 23 (72)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 4 (4) | 19 (27)
constitutional Symptoms (General disorders) | 0 (0) | 0 (0) | 4 (7) | 15 (26)
Metabolic (General disorders) | 0 (0) | 0 (0) | 3 (3) | 12 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-07-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT00634634/Prot_SAP_000.pdf
  • Informed Consent Form (2013-02-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT00634634/ICF_001.pdf